CLINICAL TRIAL: NCT00381810
Title: An Open-label, Single-arm, Multicenter Phase II/III Extension Study to Evaluate the Safety of Rituximab Re-treatment in Subjects With Moderate to Severe Systemic Lupus Erythematosus Previously Enrolled in Protocol U2971g
Brief Title: A Study to Evaluate the Safety of Rituximab Retreatment in Subjects With Systemic Lupus Erythematosus
Acronym: VOYAGER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: During a safety review of studies U2970g and U2971g, the Data Monitoring Committee recommended that enrollment in this extension trial be terminated.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U3389g
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2009-12-18 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Rituxan; SLE; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Rituximab; Methylprednisolone; Acetaminophen; Diphenhydramine

ARMS (1):
- Rituximab 1000 mg (Experimental): Participants will receive rituximab 1000 mg intravenously twice, 14 days apart at study entry and again 6 months later. Participants will also receive methylprednisolone 100 or 125 mg IV, acetaminophen 1000 mg orally, and diphenhydramine 50 mg orally prior to study drug infusion.
  Interventions: Drug: Rituximab; Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Rituximab — Rituximab will be supplied as a liquid for intravenous infusion.
Drug: Methylprednisolone
Drug: Acetaminophen
Drug: Diphenhydramine

SUMMARY:
This is a Phase II/III open label, single-arm, multicenter, extension study to evaluate the safety and efficacy of rituximab when administered on a scheduled basis every 6 months over the course of 1 year with reassessment of response at 12 months. This study is open to participants previously enrolled in Genentech Study U2971g only.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with systemic lupus erythematosus (SLE) who participated and satisfactorily completed their Week 52 evaluation in Study U2971g.
* For partial clinical response (PCR) or nonclinical response (NCR), active disease at screening as defined by one or more domains with a British Isles Lupus Assessment Group (BILAG) A score or 2 or more domains with a BILAG B score.

Exclusion Criteria:

* Subjects who were withdrawn from study U2971g because of protocol non-compliance or for safety issues.
* Any safety concern potentially attributed to rituximab that in the investigator's opinion would jeopardize subject safety.
* Subjects who were withdrawn from study U2971g and received rituximab rescue therapy outside of the protocol.
* Subjects, that in the investigator's opinion, have not demonstrated any clinical improvement by Week 52 in study U2971g and in whom the proposed therapy would represent risk without benefit.
* Unstable subjects with thrombocytopenia experiencing or at high risk for developing clinically significant bleeding or organ dysfunction requiring therapies such as plasmapheresis or acute blood or platelet transfusions.
* Pregnant women or nursing (breastfeeding) mothers.
* History of severe, allergic, or anaphylactic reactions to humanized or murine monoclonal antibodies.
* Known active infection of any kind (excluding fungal infection of nail beds) or any major episode of infection requiring hospitalization or treatment with intravenous (IV) antibiotics within 8 weeks of screening or oral antibiotics within 2 weeks prior to screening.
* History of cancer, including solid tumors, hematological malignancies, and carcinoma in situ.
* Major surgery within 4 weeks prior to screening.
* Intolerance or contraindication to oral or IV corticosteroids.
* Positive hepatitis B surface antigen (BsAg) or hepatitis C serology.
* Receipt of a live vaccine within 28 days prior to treatment.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-06-22 (Actual); Primary Completion 2008-07-31 (Actual); Study Completion 2012-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Brunetta, M.D., Study Director — Genentech, Inc.
Locations (11):
- United States (11):
  - Arizona Arthritis & Rheumatology Research, Pllc, Paradise Valley, Arizona
  - Eden Medical Center San Leandro Hospital, San Leandro, California
  - Intermountain Research Center, Boise, Idaho
  - Coeur D'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - North Shore - Long Island Jewish Hospital Health System; Rheumatology & Allergy- Clinical Immunology, Great Neck, New York
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Medical Univ of South Carolina, Charleston, South Carolina
  - Texas Research Center, Sugar Land, Texas
  - Seattle Rheumatology Assoc; Swedish Rheumatology Research, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab 1000 mg: Participants received rituximab 1000 mg intravenously twice, 14 days apart at study entry and again 6 months later. Participants also received methylprednisolone 100 or 125 mg IV, acetaminophen 1000 mg orally, and diphenhydramine 50 mg orally prior to study drug infusion.
Period: Treatment and Safety Follow-up
Arm/Group | Rituximab 1000 mg
Started | 31
Completed | 16
Not Completed | 15
Period: B Cell Follow-up
Arm/Group | Rituximab 1000 mg
Started | 7 (Participants only entered the B cell follow-up period if their peripheral B cells were depleted.)
Completed | 0
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (12.3)
Age, Customized [Number; unit: participants]
  20-64 years | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event
Description: A serious adverse event is defined as an adverse event that results in death, is life threatening, requires hospitalization, results in significant disability, results in birth defect, or is considered a significant medical event by the investigator.
Time Frame: Baseline to the end of the study (up to 52 weeks)
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 31
Percentage of participants | 35.5

ADVERSE EVENTS:
Arm/Group | Rituximab 1000 mg
Serious Adverse Events (participants affected / at risk) | 11/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 1000 mg (N=31)
Cardiac Failure Congestive (Cardiac disorders) | 1
Angina Pectoris (Cardiac disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lobar Pneumonia (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Animal Bite (Injury, poisoning and procedural complications) | 1
Pubic Rami Fracture (Injury, poisoning and procedural complications) | 1
International Normalised Ratio Increased (Investigations) | 1
Obesity (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Cerebral Infarction (Nervous system disorders) | 1
Lupus Nephritis (Renal and urinary disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Lupus Enteritis (Gastrointestinal disorders) | 1
Megacolon (Gastrointestinal disorders) | 1
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Postoperative Wound Infection (Infections and infestations) | 1
Psuedomonal Bacteraemia (Infections and infestations) | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Heamorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 1000 mg (N=31)
Lymphopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 3
Cushingoid (Endocrine disorders) | 2
Vision Blurred (Eye disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 5
Abdominal Pain (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3
Abdominal Discomfort (Gastrointestinal disorders) | 2
Mouth Ulceration (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 2
Pain (General disorders) | 5
Chest Pain (General disorders) | 3
Fatigue (General disorders) | 5
Influenza like Illness (General disorders) | 4
Oedema Peripheral (General disorders) | 3
Pyrexia (General disorders) | 2
Adverse Drug Reaction (General disorders) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 17
Sinusitis (Infections and infestations) | 15
Urinary Tract Infection (Infections and infestations) | 11
Gastroenteritis (Infections and infestations) | 5
Candidiasis (Infections and infestations) | 4
Oral Candidiasis (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 4
Herpes Zoster (Infections and infestations) | 3
Herpes Virus Infection (Infections and infestations) | 2
Gastroenteritis Viral (Infections and infestations) | 2
Viral Pharyngitis (Infections and infestations) | 2
Fungal Infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Procedural Pain (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 3
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Headache (Nervous system disorders) | 7
Migraine (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 4
Sleep Disorder (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 5
Flushing (Vascular disorders) | 3
Raynaud's Phenomenon (Vascular disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Nodule (General disorders) | 2

LIMITATIONS AND CAVEATS:
Since study U2971g did not demonstrate efficacy, a decision was made not to evaluate efficacy in this study and only safety results were evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.